CLINICAL TRIAL: NCT05769660
Title: An Open-label, Phase I Clinical Trial to Assess the Maximum Tolerated Dose (MTD), Safety and Efficacy of BEY1107 in Combination with Temozolomide in Patient with Recurrent or Progressive Glioblastoma Multiforme (GBM)
Brief Title: A Study to Evaluate Safety and Efficacy of BEY1107 in Combination with Temozolomide in Patients with Recurrent or Progressive Glioblastoma Multiforme (GBM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeyondBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BEY-2021-02
Record Dates: First submitted 2023-02-05; First posted 2023-03-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BEY1107 + Temozolomide (Experimental): Administer BEY1107 in combination with Temozolomide, 4-weeks as 1 cycle.
  Interventions: Drug: BEY1107; Combination Product: Temozolomide

INTERVENTIONS:
Drug: BEY1107 — Administer twice daily, PO, 4-week continuous dose.
Combination Product: Temozolomide — Administer once daily, PO, 5-day continuous dose, followed by 23-day rest period.

SUMMARY:
This is a Phase 1 study to evaluate the maximum tolerated dose, safety and efficacy of BEY1107 in combination with Temozolomide in Patients with Recurrent or Progressive Glioblastoma Multiforme (GBM)

DETAILED DESCRIPTION:
In Phase 1, patients with recurrent or progressive glioblastoma multiforme who failed with the standard of care will be enrolled at each dose level of BEY1107 in combination with Temozolomide.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged over 19 years or older at the time of Informed Consent.
2. Diagnosed with GBM according to the World Health Organization(WHO) criteria.
3. Subjects with progression or recurrence, with no response to the initial standard of care after being confirmed as GBM on histopathology.
4. Subjects with 1 or more lesions that are measurable or evaluable according to the Response Assessment in Neuro-Oncology(RANO) criteria.
5. Subjects with European Cooperative Oncology Group(ECOG) performance status 0 or 1.
6. For Subjects using corticosteroids, those who do not need escalation within at least 2 weeks prior to administration of Investigational Product(IP) and on a stable dose.
7. Women of childbearing potential who are not surgically sterile must consent to practice acceptable contraception until 6 months after the end of IP administration and also have the evidence of not being fertile.

8 Non-vasectomized men who consent to use an acceptable contraception by one-self and the partner until 3 months after the end of IP administration.

9. Subjects who are fully informed of this trial, voluntarily decide to participate in the trial and provide written consent to comply with requirements for the trial.

Exclusion Criteria:

1. Patients with a history of chemotherapy for treatment of recurrent glioblastoma multiforme after the initial standard of care as of screening.
2. Subjects who have not recovered from the toxicity of the prior anticancer therapy.
3. Subjects who have past history of major gastrointestinal surgery making oral drug administration impossible or possibly affecting absorption of IP.
4. Subjects who had a major surgery requiring general anesthesia within 4 weeks of screening.
5. Subjects with a history of other malignancy except adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ, papillary thyroid cancer or early gastric cancer.
6. Subjects with a genetic problem(eg. Galactose intolerance).
7. Subjects with hypersensitivity to the ingredient(s) or excipient(s) of the investigational product (BEY1107) or temozolomide.
8. Subjects with hypersensitivity to dacarbazine (DTIC).
9. Subjects who have the cardiovascular disease as of screening.
10. Active hepatitis B, C or HIV positive.
11. Patients with acute or severe infection.
12. Subjects who take a Rifampin, Phenytoin and azole class antifungal drugs in combination.
13. Subjects who had been administered other IP within 4 weeks prior to screening.
14. Patients with inadequate bone marrow, kidney and liver function.
15. Pregnant women, breastfeeding women, or positive findings on the pregnancy test at screening.
16. Subjects with life expectancy of less than 12 weeks by the investigator.
17. Subjects determined by the investigator to be ineligible for participation in this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | From baseline up to disease progression, approximately 4 weeks
  MTD will be assessed based on dose-limiting toxicity(DLT) assessment
Recommended Phase II Dose (RP2D) assessed by investigator following administration of BEY1107 in combination with Temozolomide in Phase I. | From baseline up to disease progression, approximately 48 weeks
  RP2D will be assessed based on MTD.

SECONDARY OUTCOMES:
Disease control rate(DCR) | From baseline up to disease progression, approximately 48 weeks
  DCR is defined as the proportion of participants who achieved a confirmed best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD)
Progression-free survival(PFS) rate at 6 months | From baseline up to 6 months
  PFS is defined as the time from the start of study treatment to the date of the first documentation of objective progressive disease(PD) or death due to any cause, whichever is earlier
Pharmacokinetic(PK) of maximum serum Concentration (Cmax) | From baseline up to 4 weeks post-dose
  Plasma concentrations at each time point and PK parameters Cmax of BEY1107 will be assessed in the PK sampling cohort
Pharmacokinetic of Time to Reach Maximum Serum Concentration (Tmax) | From baseline up to 4 weeks post-dose
  Plasma concentrations at each time point and PK parameters Tmax of BEY1107 will be assessed in the PK sampling cohort
Pharmacokinetic of Area Under the Serum Concentration-Time Curve Up to Last Quantifiable Time (AUClast) | From baseline up to 4 weeks post-dose
  Plasma concentrations at each time point and PK parameters AUC last of BEY1107 will be assessed in the PK sampling cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No